CLINICAL TRIAL: NCT00321997
Title: A PHASE II/III RANDOMIZED, DOUBLE-MASKED, CONTROLLED, DOSE-RANGING, MULTI-CENTER COMPARATIVE TRIAL, IN PARALLEL GROUPS, TO ESTABLISH THE SAFETY AND EFFICACY OF INTRAVITREAL INJECTIONS OF EYE001 (ANTI-VEGF PEGYLATED APTAMER) GIVEN EVERY 6 WEEKS FOR 54 WEEKS, IN PATIENTS WITH EXUDATIVE AGE-RELATED MACULAR DEGENERATION (AMD)
Brief Title: A Clinical Trial to Explore Safety and Efficacy of Different Doses of Pegaptanib Sodium, Compared to Sham, in Patients With Wet AMD.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eyetech Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOP1003 and EOP1004
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Last update posted 2006-05-04 (Estimated); Status verified 2006-05

CONDITIONS: Age-Related Macular Degeneration
Keywords: AMD; Age-Related Macular Degeneration; Macular Degeneration; Macugen; pegaptanib sodium
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

INTERVENTIONS:
Drug: Pegaptanib sodium

SUMMARY:
The purpose of this study is to compare the ability of different doses of pegaptanib sodium to safely and effectively minimize fluid leakage within the eye, thereby stabilizing or impriving vision in patients with wet AMD when compared to placebo injections.

ELIGIBILITY:
Inclusion Criteria:

Subjects of either gender, aged 50 years or greater. Subfoveal choroidal neovascularization (CNV) due to AMD. Best corrected visual acuity in the study eye between 20/40 and 20/320.

Exclusion Criteria:

Any prior subfoveal thermal laser therapy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540
Dates: Start 2001-05; Study Completion 2007-10

REFERENCES:
- [Derived] Boyer DS, Goldbaum M, Leys AM, Starita C; V.I.S.I.O.N. Study Group. Effect of pegaptanib sodium 0.3 mg intravitreal injections (Macugen) in intraocular pressure: posthoc analysis from V.I.S.I.O.N. study. Br J Ophthalmol. 2014 Nov;98(11):1543-6. doi: 10.1136/bjophthalmol-2013-304075. Epub 2014 Jul 4. PMID 24997182